CLINICAL TRIAL: NCT03196349
Title: Comparison of Oral Anticoagulants for Extended VEnous Thromboembolism (COVET)
Brief Title: Comparison of Oral Anticoagulants for Extended VEnous Thromboembolism
Acronym: COVET
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Duke University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00077510
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2019-08-14 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Warfarin; apixaban; Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Warfarin (Active Comparator): Subjects randomized to Warfarin will have warfarin administered daily in order to maintain a target INR of 2-3
  Interventions: Drug: Warfarin
- Apixaban (Active Comparator): Subjects randomized to Apixaban will have apixaban administered study drug of 2.5mg twice daily
  Interventions: Drug: Apixaban 2.5 MG
- Rivaroxaban (Active Comparator): Subjects randomized to Rivaroxaban will have rivaroxaban administered study drug of 10 mg daily
  Interventions: Drug: Rivaroxaban 10 MG

INTERVENTIONS:
Drug: Warfarin — Will be randomized to receive open label warfarin daily to achieve a target INR of 2-3
  Arms: Warfarin
Drug: Apixaban 2.5 MG — Will be randomized to receive open label apixaban of 2.5 mg twice daily
  Arms: Apixaban
Drug: Rivaroxaban 10 MG — Will be randomized to receive open label rivaroxaban of 10mg daily
  Arms: Rivaroxaban

SUMMARY:
Comparison of Oral anticoagulants (warfarin, apixaban and rivaroxaban) for extended VEnous Thromboembolism.

DETAILED DESCRIPTION:
Determine if apixaban is superior to warfarin in the reduction of clinically relevant bleeding. Determine if rivaroxaban is superior to warfarin in the reduction of clinically relevant bleeding. Determine if apixaban is non-inferior to warfarin in the prevention of recurrent venous thromboembolism. Determine if rivaroxaban is non-inferior to warfarin in the prevention of recurrent venous thromboembolism. An exploratory comparison of apixaban versus rivaroxaban for the prevention of clinically relevant bleeding and recurrent Venous Thromboembolism (VTEs) as a secondary objective.

ELIGIBILITY:
3.1 Inclusion Criteria

To be eligible for this trial, patients must meet all of the following criteria:

* Have confirmed acute, symptomatic, first lower extremity proximal DVT and/or PE that is NOT associated with a transient risk factor.
* Have completed an initial treatment course of oral anticoagulant therapy for 3-12 months and have a recommendation from their provider to continue anticoagulation indefinitely.
* Have the capacity to understand and sign an informed consent form.
* Be 18 years of age and older.
* Under the direct care of a healthcare provider for treatment of VTE for the length of time in the study.

3.2 Exclusion Criteria

If a patient meets any of the following criteria, he or she may not be enrolled in the study:

* Creatinine clearance (CrCl) < 30 mL/min as determined by Cockcroft-Gault formula documented within 3 months from date of consent
* Significant liver disease (Child-Pugh B or C)
* Concomitant use of medications that are strong P-glycoprotein or CYP3A4 inducers/inhibitors
* Another indication for chronic therapeutic-dose anticoagulation, such as atrial fibrillation (i.e., rivaroxaban, 10 mg daily, or apixaban, 2.5 mg twice daily, would not be appropriate therapy)
* A clinical indication for a specific anticoagulant regimen (e.g., warfarin with a target INR of 2-3 is recommended for patients with 'triple-positive' antiphospholipid syndrome).
* Life expectancy < 3 months
* Currently pregnant or breast feeding
* Unable / unwilling to pay for one (or more) of the treatment options
* Active Cancer defined as:

Diagnosed with cancer within the past 6 months; or Recurrent, regionally advanced or metastatic disease; Currently receiving treatment or have received any treatment for cancer during the 6 months prior to randomization; or A hematologic malignancy not in complete remission

• Unwilling / unlikely to agree to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ortel, MD, Principal Investigator — Duke University
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Started | 17 | 14 | 13
Completed | 0 | 0 | 0
Not Completed | 17 | 14 | 13
Not completed — Did not receive study drug | 0 | 1 | 2
Not completed — No data entered | 2 | 4 | 0
Not completed — Study Terminated early | 15 | 9 | 11

BASELINE CHARACTERISTICS:
Population: 44 subjects were randomized yet only 31 were on study drug by the 1 month telephone follow up. Due to the study being stopped early some of the data was outstanding in the database which is why the numbers do not add up to 44 in all of the categories.
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin | Apixaban | Rivaroxaban | Total
Number analyzed (Participants) | 16 | 13 | 12 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 5 | 11 | 27
  >=65 years | 5 | 8 | 1 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 12 | 10 | 10 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: In the Apixaban arm 1 subject was never administered study drug and in the rivaroxaban 2 subjects never received study drug. They were excluded from the analysis.
  Participants
    number analyzed (Participants) | 16 | 12 | 11 | 39
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 1 | 2 | 5
    White | 14 | 10 | 8 | 32
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 7 | 9 | 26
  Canada | 6 | 6 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinically Relevant Bleeding Events
Description: Primary outcome of Clinically relevant bleeding (composite of major bleeding (MB) and/or clinically relevant non major bleeding (CRNMB))
Time Frame: Randomization to 12 months
Population: 44 subjects were randomized but analysis was only done on participants that had started therapy by the 1 month telephone visit
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Number analyzed (Participants) | 14 | 8 | 9
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Recurrent Venous Thromboembolism (VTE)
Description: Primary efficacy outcome of recurrent VTE
Time Frame: Randomization to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Number analyzed (Participants) | 17 | 14 | 13
Participants | 0 | 1 | 0

3. Other Pre Specified Outcome: Number of Subjects Experiencing Major Bleeding
Description: Major bleeding
Time Frame: Randomization to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Number analyzed (Participants) | 17 | 14 | 13
Participants | 0 | 0 | 0

4. Other Pre Specified Outcome: Number of Subjects Experiencing Clinically Relevant Non-major Bleeding
Description: Clinically relevant non-major bleeding
Time Frame: Randomization to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Number analyzed (Participants) | 17 | 14 | 13
Participants | 0 | 0 | 0

5. Other Pre Specified Outcome: Number of Subjects With Premature Termination of Study Medication
Description: Premature termination of study medication
Time Frame: Randomization to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Number analyzed (Participants) | 17 | 14 | 13
Participants | 0 | 0 | 0

6. Other Pre Specified Outcome: Number of Subjects Experiencing All-cause Mortality
Description: All cause mortality
Time Frame: Randomization to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Number analyzed (Participants) | 17 | 14 | 13
Participants | 0 | 0 | 0

7. Other Pre Specified Outcome: Number of Subjects Experiencing Vascular Events (Myocardial Infarction, Ischemic Stroke)
Description: MI, ischemic stroke, peripheral arterial embolism
Time Frame: Randomization to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin | Apixaban | Rivaroxaban
Number analyzed (Participants) | 17 | 14 | 13
Participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 9 months
Arm/Group | Warfarin | Apixaban | Rivaroxaban
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03196349/SAP_002.pdf
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03196349/Prot_003.pdf
  • Informed Consent Form (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT03196349/ICF_004.pdf